CLINICAL TRIAL: NCT03697473
Title: A Comparison of Hip Extension and Nordic Hamstring Exercise Programmes on Isokinetic Hamstring Strength
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dublin City University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2016_007_EW
Record Dates: First submitted 2018-09-27; First posted 2018-10-05 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Hamstring Injury
Keywords: Hamstring strength; Isokinetics; Nordic hamstring exercise; Eccentric strength; Hip extension exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The principal investigator responsible for the statistical analysis was blinded to the group allocation of participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nordic Hamstring Exercise Group (Active Comparator): Participants were required to kneel on a gym mat keeping their hips in a slightly flexed position and to slowly lower themselves in a controlled manner as far as they could towards the ground. When they could no longer lower themselves as such, they were instructed to utilise their arms to buffer the fall and touch their chest off the ground, while maintaining tension in their hamstrings. Once their chest touched the ground they were instructed to immediately return to the starting position by pushing up with their hands.
  Interventions: Other: Nordic hamstring exercise
- Hip Extension Exercise Group (Experimental): The participant lay on an exercise bench at a 45° angle with their hips held just over the top of the bench, their trunk erect and hips extended and their heel supported. Participants slowly flexed their hip until they reached 90° from the starting position and were then required to return to the starting position by extending through the hip while maintaining a neutral pelvic and trunk posture throughout. This exercise was then repeated on the opposite leg
  Interventions: Other: Hip extension exercise

INTERVENTIONS:
Other: Nordic hamstring exercise — The exercise protocol consisted of the following sets and repetitions Week 1 - 2 sessions with 2 sets of 6 repetitions. Week 2 - 2 sessions with 3 sets of 6 repetitions Week 3 - 2 sessions with 4 sets of 8 repetitions. Week 4 - 2 sessions with 4 sets of 10 repetitions.
  Arms: Nordic Hamstring Exercise Group
Other: Hip extension exercise — The exercise protocol consisted of the following sets and repetitions Week 1 - 2 sessions with 2 sets of 6 repetitions. Week 2 - 2 sessions with 3 sets of 6 repetitions Week 3 - 2 sessions with 4 sets of 8 repetitions. Week 4 - 2 sessions with 4 sets of 10 repetitions.
  Arms: Hip Extension Exercise Group

SUMMARY:
This study aimed to compare the effect of two hamstring strengthening programmes on hamstring muscle strength in Gaelic footballers. 26 Gaelic footballers were recruited and randomly assigned to one of two 4-week hamstring strengthening programmes, namely the hip extension exercise programme and the Nordic hamstring exercise protocol. Isokinetic hamstring and quadriceps strength were measured before and after the intervention.

DETAILED DESCRIPTION:
Recruitment:

Participants were recruited from the local university sports clubs. Club chairpersons were asked to send an email to club players. Players interested in participating in the study expressed an interest by replying to the email. Potential participants were asked to attend a meeting where they had the study explained to them. Those who were interested were then assessed for inclusion and exclusion criteria.

Group allocation:

A four block randomisation method was used to allocate participants to the Nordic hamstring exercise protocol or the hip extension exercise protocol.

Interventions:

The Nordic hamstring exercise protocol or the hip extension exercise protocol

Testing procedure:

The isokinetic strength of the participants' hamstrings and quadriceps were recorded before and after the exercise intervention.

A 10 point visual analogue scale was used to record the level of muscle soreness experienced after each training session.

ELIGIBILITY:
Inclusion Criteria:

* male
* free from hamstring injury in the 6 months prior to the study
* currently playing Gaelic football at a varsity level on at least three occasions per week

Exclusion Criteria:

* history of a hip or knee injury in the 3 months prior to the study
* a history of anterior cruciate ligament rupture
* a history of involvement in a hamstring strengthening, injury prevention programme in the 3 months prior to the study.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2017-01-05 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Peak isokinetic eccentric hamstring strength at 60°.s-1 | Change from baseline assessment at six weeks
  This was measured using an isokinetic dynamometer

SECONDARY OUTCOMES:
Functional hamstring-to-quadriceps ratio at 60°.s-1 | Change from baseline assessment at six weeks
  This was calculated by dividing the peak isokinetic, eccentric hamstring strength at 60°.s-1 by the peak isokinetic, concentric quadriceps strength at 60°.s-1
Between limb, isokinetic eccentric hamstring strength asymmetries | Change from baseline assessment at six weeks
  Between limb eccentric strength percentage asymmetries were calculated as a non-dominant/dominant ratio converted to percentage difference using log transformation.
Muscle soreness rating following exercise | 1 minute at the end of each intervention session
  Participants used a 10 point visual analogue scale to record the level of muscle soreness experienced after training sessions.
  The scale consisted of a single scale of 0 to 10 where 0 was no soreness at all and 10 was the greatest soreness they could imagine. A higher score indicated a worse outcome. There are no subscales included in this.

CONTACTS AND LOCATIONS:
Overall Officials: Enda Whyte, PhD, Principal Investigator — Dublin City University; Siobhán O'Connor, PhD, Principal Investigator — Dublin City University

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised data may be shared to allow future analysis by other researchers

REFERENCES:
- [Background] van der Horst N, Smits DW, Petersen J, Goedhart EA, Backx FJ. The preventive effect of the nordic hamstring exercise on hamstring injuries in amateur soccer players: a randomized controlled trial. Am J Sports Med. 2015 Jun;43(6):1316-23. doi: 10.1177/0363546515574057. Epub 2015 Mar 20. PMID 25794868
- [Background] Bourne MN, Timmins RG, Opar DA, Pizzari T, Ruddy JD, Sims C, Williams MD, Shield AJ. An Evidence-Based Framework for Strengthening Exercises to Prevent Hamstring Injury. Sports Med. 2018 Feb;48(2):251-267. doi: 10.1007/s40279-017-0796-x. PMID 29116573
- [Background] Bourne MN, Duhig SJ, Timmins RG, Williams MD, Opar DA, Al Najjar A, Kerr GK, Shield AJ. Impact of the Nordic hamstring and hip extension exercises on hamstring architecture and morphology: implications for injury prevention. Br J Sports Med. 2017 Mar;51(5):469-477. doi: 10.1136/bjsports-2016-096130. Epub 2016 Sep 22. PMID 27660368
- [Background] Bijur PE, Silver W, Gallagher EJ. Reliability of the visual analog scale for measurement of acute pain. Acad Emerg Med. 2001 Dec;8(12):1153-7. doi: 10.1111/j.1553-2712.2001.tb01132.x. PMID 11733293
- [Background] Impellizzeri FM, Bizzini M, Rampinini E, Cereda F, Maffiuletti NA. Reliability of isokinetic strength imbalance ratios measured using the Cybex NORM dynamometer. Clin Physiol Funct Imaging. 2008 Mar;28(2):113-9. doi: 10.1111/j.1475-097X.2007.00786.x. Epub 2007 Dec 7. PMID 18070123
- [Background] Lee JWY, Mok KM, Chan HCK, Yung PSH, Chan KM. Eccentric hamstring strength deficit and poor hamstring-to-quadriceps ratio are risk factors for hamstring strain injury in football: A prospective study of 146 professional players. J Sci Med Sport. 2018 Aug;21(8):789-793. doi: 10.1016/j.jsams.2017.11.017. Epub 2017 Dec 5. PMID 29233665
- [Background] Opar DA, Williams MD, Timmins RG, Hickey J, Duhig SJ, Shield AJ. Eccentric hamstring strength and hamstring injury risk in Australian footballers. Med Sci Sports Exerc. 2015 Apr;47(4):857-65. doi: 10.1249/MSS.0000000000000465. PMID 25137368
- [Derived] Whyte EF, Heneghan B, Feely K, Moran KA, O'Connor S. The Effect of Hip Extension and Nordic Hamstring Exercise Protocols on Hamstring Strength: A Randomized Controlled Trial. J Strength Cond Res. 2021 Oct 1;35(10):2682-2689. doi: 10.1519/JSC.0000000000003220. PMID 31356512